CLINICAL TRIAL: NCT04654039
Title: Post-Marketing Surveillance (PMS) Protocol of REKOVELLE Pre-Filled Pen(Follitropin Delta)
Brief Title: Post-Marketing Surveillance (PMS) Protocol of REKOVELLE Pre-Filled Pen (Follitropin Delta)
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000385
Record Dates: First submitted 2020-11-16; First posted 2020-12-04 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Infertility, Female
Keywords: Follitropin Delta; REKOVELLE
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment of Infertility: Non intervention
  Interventions: Other: Other: Non intervention

INTERVENTIONS:
Other: Other: Non intervention — Non intervention

SUMMARY:
This post-marketing surveillance study was conducted in accordance with the regulations for re-examination of domestic new drugs (Standard for Re-Examination of New Drugs: Ministry of Food and Drug Safety [MFDS]: Notification No. 2017-95, 21 Nov, 2017).

It was important to monitor the pattern of drug use in general practice for a long term after marketing authorization, and to investigate and identify potential new adverse events (AEs) and their onset status that were not observed during the drug development phases and any potential factors that affect safety and effectiveness of the new drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were prescribed with REKOVELLE (follitropin delta) for the first time according to the approved administration method and dose
* Participants who have consented to personal information use

Exclusion Criteria:

* Participants who are prohibited from use according to the special warnings and precautions for use of REKOVELLE (follitropin delta)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Participants receiving REKOVELLE pre-filled pen (follitropin delta) within the range of the approved product labeling in Korea. Participants were enrolled only after the treatment decision had been made and no aspect of this study would interfere with or influence the routine medical procedures and/or medications received.
Sampling Method: Probability Sample
Enrollment: 728 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with serious AEs and adverse drug reactions (ADRs) | Until the 10 to 11 weeks after the embryo transfer or until the 30 days after treatment termination
Proportion of subjects with unexpected AEs/ADRs not reflected in 'Precautions for Use' | Until the 10 to 11 weeks after the embryo transfer or until the 30 days after treatment termination
Proportion of subjects with expected ADRs | Until the 10 to 11 weeks after the embryo transfer or until the 30 days after treatment termination
Proportion of subjects with non-serious ADRs | Until the 10 to 11 weeks after the embryo transfer or until the 30 days after treatment termination
Proportion of subjects with ovarian hyperstimulation syndrome (OHSS) | Until the 10 to 11 weeks after the embryo transfer or until the 30 days after treatment termination
Technical malfunction of REKOVELLE pre-filled pen | Until the 10 to 11 weeks after the embryo transfer or until the 30 days after treatment termination

SECONDARY OUTCOMES:
Number of the oocytes retrieved | At the oocyte retrieval visit, after completion of controlled ovarian stimulation and approximately 36 hours after human chorionic gonadotropin (hCG) administration.
Ongoing pregnancy rate in women undergoing controlled ovarian stimulation | Between 10-11 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (15):
- South Korea (15):
  - Pyeongchon Maria, 8/9F, Olympic Sports Center120, Dongan-ro, Dongan-gu, Anyang
  - Dream-I clinic, 45-17, Huimang-ro 46beon-gil, Baebang-eup, Asan
  - Centum Eroom Woman Clinic, 10F, Centum Tower Medical, 20, Centum-2-ro, Haeundae-gu, Busan
  - Eroom women's clinic, 25, Seomyeon-ro, Busanjin-gu, Busan
  - Seoul Women's Hospital, 7, Munjeong-ro, Seo-gu, Daejeon
  - Creation And Love Women's Hospital, 957, Mujin-daero, Seo-gu, Gwangju
  - Mirae and Heemang Women's Hospital, 7F, Dana Medical Center, 68, Jukbong-daero, Seo-gu, Gwangju
  - Design Hospital, Jeonju
  - Trinium Woman's Hospital, 1834, MainTower, Hannuridae-ro, Sejong
  - CHA university Bundang medical center, 59, Yatap-ro, Bundang-gu, Seongnam
  - Seoul Nation University Bundang Hospital, 82, Gumi-ro 173beon-gil, Bundang-gu, Seongnam
  - M Fertility Center, 12F, 407, Teheran-ro, Gangnam-gu, Seoul
  - MariaS (Sangbong), 267, Mangu-ro, Jungnang-gu, Seoul
  - Mizmedi Hospital, 295, Gangseo-ro, Gangseo-gu, Seoul
  - Seoul Maria Fertility Hospital, 20, Cheonho-daero, Dongdaemun-gu, Seoul